CLINICAL TRIAL: NCT00210665
Title: A Multicenter, Open-Label, Single-Arm Study of YONDELIS (Trabectedin) for Subjects With Locally Advanced or Metastatic Soft Tissue Sarcoma Who Have Relapsed or Are Refractory to Standard of Care Treatment
Brief Title: A Study to Provide Access to Trabectedin in Participants With Locally Advanced or Metastatic Soft Tissue Sarcoma Who Have Persistent or Recurrent Disease and Who Are Not Expected to Benefit From Currently Available Standard of Care Treatment
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR003583; ET743SAR3002 (Other: Janssen Research & Development, LLC); NCT00707109 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Sarcoma
Keywords: Sarcoma; Soft tissue sarcoma; Standard care; Trabectedin; Antitumor agent; Safety
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Type= exact number, unit= mg/m2, number= 1.5, form= intravenous infusion, route= intravenous use. 1.5mg/m2 as 24hr infusion on day 1 of each 21 day cycle

SUMMARY:
The purpose of this study is to facilitate access to trabectedin for eligible previously treated patients with soft tissue sarcoma (STS), who cannot be expected to benefit from currently available therapeutic options but who may benefit from treatment with trabectedin. The safety profile of trabectedin will be evaluated to further assess the potential risks of trabectedin treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label (all people know the identity of the intervention), single-arm study. It will consist of 2 Phases: a Screening Phase (up to 21 days before the first dose administration), and Treatment Phase (for patients meeting the continuation criteria). During the Treatment Phase, patients will receive a dose of 1.5 mg/m2 trabectedin intravenous formulation administered as a 24-hour infusion on Day 1 of each suggested 21-day treatment cycle. All patients will receive 20 mg dexamethasone (or corticosteroid equivalent to dexamethasone). Number of cycles is not specified for this study. Patients may continue to receive treatment as long as they obtain an overall clinical benefit, ie, until there is clear evidence of disease progression or unacceptable toxicity, as judged by the investigator. Trabectedin is the first of a new class of antitumor agents. Previous studies with trabectedin in patients who had been previously treated for soft tissue sarcoma have suggested that treatment with trabectedin resulted in tumor shrinkage, disease stabilization, and improved survival rates. However, hematologic toxicity, hepatic toxicity, and renal impairment were also observed in these patients. The safety profile of trabectedin will be evaluated to further assess the potential risks of trabectedin treatment in patients previously treated for soft tissue sarcoma who are not expected to benefit from currently available therapeutic options for treatment of soft tissue sarcoma. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable advanced or metastatic histologically proven soft tissue sarcoma (STS). Eligibility will include adult participants with desmoplastic small round cell tumor
* Must have relapsed or had progressive disease following standard of care treatment with chemotherapy prior to enrollment or intolerant to prior standard of care treatment with chemotherapy due to safety issues
* Recovery from toxic effects of prior therapies to Grade 1 or better according to National Cancer Institute-Common Terminology Criteria of Adverse Events (criteria used to grade the severity of toxic effects on a scale from 0 to 5 - Grade 1 = mild in severity, Grade 0 = no severity)
* Clinical test results within acceptable limits (ie, hematologic, clinical chemistry and hepatic function test results)
* Female participants must be postmenopausal, surgically sterile, abstinent, or if sexually active, be practicing 2 effective methods of birth control (eg, prescription hormonal contraceptive, intrauterine device, double-barrier method [eg, condoms, occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, cream, gel, film, or suppository]), before entry, and must agree to continue to use these same methods of contraception throughout the study and for 3 months thereafter. Male participants must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm for a minimum of 5 months after treatment discontinuation

Exclusion Criteria:

* Diagnosis of Ewing's sarcoma or osteosarcoma, less than 3 weeks from last dose of radiation, systemic cytotoxic therapy (or 4 half lives, whichever is longer)
* Active symptomatic viral hepatitis or chronic liver disease
* Significant uncontrolled cardiac condition, including New York Heart Association Class II or greater heart failure, uncontrolled angina pectoris, myocardial infarction within 6 months before enrollment, significant pericardial disease, or uncontrolled or arrhythmias
* Active infection
* Female participant who is pregnant or breastfeeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC & Development, L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (36):
- United States (31):
  - Anchorage, Alaska
  - San Diego, California
  - Santa Monica, California
  - Aurora, Colorado
  - Daytona Beach, Florida
  - Hollywood, Florida
  - Atlanta, Georgia
  - Coeur d'Alene, Idaho
  - Park Ridge, Illinois
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - Saint Joseph, Missouri
  - Omaha, Nebraska
  - Newark, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (4):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
  - Edmonton
- Tel Aviv, Israel

REFERENCES:
- [Derived] Samuels BL, Chawla S, Patel S, von Mehren M, Hamm J, Kaiser PE, Schuetze S, Li J, Aymes A, Demetri GD. Clinical outcomes and safety with trabectedin therapy in patients with advanced soft tissue sarcomas following failure of prior chemotherapy: results of a worldwide expanded access program study. Ann Oncol. 2013 Jun;24(6):1703-9. doi: 10.1093/annonc/mds659. Epub 2013 Feb 5. PMID 23385197
- [Derived] Charytonowicz E, Terry M, Coakley K, Telis L, Remotti F, Cordon-Cardo C, Taub RN, Matushansky I. PPARgamma agonists enhance ET-743-induced adipogenic differentiation in a transgenic mouse model of myxoid round cell liposarcoma. J Clin Invest. 2012 Mar;122(3):886-98. doi: 10.1172/JCI60015. Epub 2012 Feb 1. PMID 22293175
- See also: A Multicenter, Open-Label Single-Arm Study of YONDELIS (trabectedin) for Subjects With Locally Advanced or Metastatic Soft Tissue Sarcoma Who Have Relapsed or are Refractory to Standard of Care Treatment — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=531&filename=CR003583_CSR_.pdf